CLINICAL TRIAL: NCT06135207
Title: The Correlation Between COVID-19 and Dysphagia in Adults With Swallowing Disorders
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Gökhan Can TÖRPÜ, Principal Investigator, Bezmialem Vakif University
Other Study IDs: BezmialemVU-GCT-02
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Dysphagia
Keywords: COVID-19; Dysphagia; Flexible endoscopic swallowing study; Oral motor dysfunction
MeSH Terms: conditions — COVID-19; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Group: Patients with a history of COVID-19 infection and experiencing symptoms of dysphagia.
- Non-COVID-19 Group: Patients who do not have a history of COVID-19 infection but experience symptoms of dysphagia.

SUMMARY:
This study aims to investigate the correlation between COVID-19 and dysphagia in adults. The population of the study consisted of those who applied to Bezmialem University, Department of Otorhinolaryngology, Dysphagia Outpatient Clinic with the complaint of dysphagia. Patients older than 18 years of age, suffering from dysphagia and not having mental retardation were included in the study. Patients who did not have swallowing difficulties and refused to participate in the study were excluded.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is characterized by involvement in multiple tissues and organs throughout the body. Conditions related to COVID-19 itself or its treatment are known to be associated with swallowing function. Our study aimed to investigate the correlation between COVID-19 and dysphagia in adults who applied to our dysphagia outpatient clinic. Patients over the age of 18, who applied to the dysphagia outpatient clinic were included in our study. Patients' demographic and COVID-19 information were recorded. Swallowing impairment of the patients was evaluated with the fiberoptic endoscopic swallowing study (FEES). FEES was scored with the Penetration-Aspiration Scale (PAS). Eating Assessment Tool-10 (EAT-10) questionnaire was used to examine how the quality of life of the patients was affected by swallowing difficulties. Oral motor dysfunction (OMD) evaluation was performed by the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Suffering from dysphagia
* Not having mental retardation

Exclusion Criteria:

* Patients who did not have swallowing difficulties
* Refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18, who applied to the dysphagia outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-10-23 (Actual)

PRIMARY OUTCOMES:
Flexible Endoscopic Evaluation of Swallowing (FEES) | Three Months
  Swallowing disorders of the patients were evaluated with fiberoptic endoscopic swallowing study (FEES).
The Penetration - Aspiration Scale | Three Months
  The results of FEES was scored by the Penetration-Aspiration Scale. The Penetration - Aspiration Scale is an 8-point scale during instrumental swallowing assessments such as the fiberoptic endoscopic swallow study, both indicating the localization of the airway leak and demonstrating the response to the assessment.
Oral Motor Dysfunction (OMD) | Three Months
  Oral motor dysfunction (OMD) assessment of the patients was performed by physical examination of the oropharyngeal mechanism. Lips, tongue, palate, cheeks, teeth, jaw, larynx, and oral reflexes were evaluated with 26 items in terms of lifting, pressing, extending, retraction, approximation, rolling, lateralization, movement, coordination, speed, tone, and strength. A scale of 1-4 was used for scoring (1=within functional limits, 2=mild impairment, 3=moderate impairment, 4=severe impairment). The total score ranged from 26 to 104, with higher scores indicating greater degree of impairment. Only a score of 26 was considered normal within functional limits.
Cranial Nerve Examination | Three Months
  Nervus trigeminus (V. cranial nerve), Nervus facialis (VII. cranial nerve), Nervus glossopharyngeus (IX. cranial nerve), Nervus vagus (X. cranial nerve) and Nervus hypoglossus (XII. cranial nerve) which are five cranial nerves involved in swallowing function were evaluated by the clinician.
Eating Assessment Tool-10 (EAT-10) | Three Months
  The Eating Assessment Tool-10 (EAT-10) was used to examine how the quality of life of the patients was affected because of their difficulty in swallowing.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan C Törpü, BPT, Principal Investigator — Bezmialem Vakif University; Müberra Tanrıverdi, PhD, Study Director — Bezmialem Vakif University; Nahide Öztoprak, BPT, Study Chair — Bezmialem Vakif University; Ömer F Çalım, PhD, Study Chair — Bezmialem Vakif University; Orhan Özturan, PhD, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vergara J, Lirani-Silva C, Brodsky MB, Miles A, Clave P, Nascimento W, Mourao LF. Potential Influence of Olfactory, Gustatory, and Pharyngolaryngeal Sensory Dysfunctions on Swallowing Physiology in COVID-19. Otolaryngol Head Neck Surg. 2021 Jun;164(6):1134-1135. doi: 10.1177/0194599820972680. Epub 2020 Nov 10. PMID 33167752
- [Background] Dziewas R, Warnecke T, Zurcher P, Schefold JC. Dysphagia in COVID-19 -multilevel damage to the swallowing network? Eur J Neurol. 2020 Sep;27(9):e46-e47. doi: 10.1111/ene.14367. Epub 2020 Jun 13. No abstract available. PMID 32460415
- [Background] Cheney DM, Siddiqui MT, Litts JK, Kuhn MA, Belafsky PC. The Ability of the 10-Item Eating Assessment Tool (EAT-10) to Predict Aspiration Risk in Persons With Dysphagia. Ann Otol Rhinol Laryngol. 2015 May;124(5):351-4. doi: 10.1177/0003489414558107. Epub 2014 Oct 30. PMID 25358607